CLINICAL TRIAL: NCT06076694
Title: Single-center, Randomized, Open-label Phase Ic/IIb Clinical Study to Evaluate the Efficacy and Safety of TNP-2198 Capsules, Rabeprazole Sodium Enteric-coated Tablets and Amoxicillin Capsules Combined With Multiple Doses of Rabeprazole Sodium Enteric-coated Tablets and Amoxicillin Capsules Compared With Multiple Doses of Rabeprazole Sodium Enteric-coated Tablets and Amoxicillin Capsules Combined With Multiple Doses in Helicobacter Pylori Infection-positive Population
Brief Title: Efficacy and Safety After Multiple Doses of TNP-2198 Capsules, Rabeprazole Sodium Enteric-coated Tablets and Amoxicillin Capsules in Helicobacter Pylori Infected-positive Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TenNor Therapeutics (Suzhou) Limited (Industry)
Responsible Party: Sponsor
Organization: TenNor Therapeutics Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNP-2198-06
Record Dates: First submitted 2023-09-26; First posted 2023-10-11 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-10

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Rabeprazole; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group A (Experimental): TNP-2198 capsules 400 mg + rabeprazole sodium enteric-coated tablets 20 mg + amoxicillin capsules 1 g; Twice daily (BID) for 14 days
  Interventions: Drug: TNP-2198; Drug: Rabeprazole Sodium; Drug: Amoxicillin
- Group B (Experimental): TNP-2198 capsules 600 mg + rabeprazole sodium enteric-coated tablets 20 mg + amoxicillin capsules 1 g; BID for 14 days
  Interventions: Drug: TNP-2198; Drug: Rabeprazole Sodium; Drug: Amoxicillin
- Group C (Experimental): TNP-2198 capsule 600 mg + rabeprazole sodium enteric-coated tablets 20 mg; Three times daily (TID) for 14 days
  Interventions: Drug: TNP-2198; Drug: Rabeprazole Sodium
- Group D (Experimental): TNP-2198 capsules 600 mg + rabeprazole sodium enteric-coated tablets 20 mg + amoxicillin capsules 1g; TID for 7 days
  Interventions: Drug: TNP-2198; Drug: Rabeprazole Sodium; Drug: Amoxicillin
- Control group (Active Comparator): Rabeprazole sodium enteric-coated tablets 20 mg + amoxicillin capsules 1 g
  Interventions: Drug: Rabeprazole Sodium; Drug: Amoxicillin

INTERVENTIONS:
Drug: TNP-2198 — Group A, TNP-2198 capsules 400mg(4 capsules),BID, 14days Group B, TNP-2198 capsules 600mg(6 capsules),BID, 14days Group C , TNP-2198 capsules 600mg(6 capsules),TID, 14days Group D, TNP-2198 capsules 600mg(6 capsules),TID, 7days
  Other Names: Rifasutenizol
  Arms: Group A; Group B; Group C; Group D
Drug: Rabeprazole Sodium — Group A,Group B,Control group: Rabeprazole sodium enteric-coated tablets 20 mg, BID, 14days Group C :Rabeprazole sodium enteric-coated tablets 20 mg, TID, 14 days Group D : Rabeprazole sodium enteric-coated tablets 20 mg, TID, 7 days
Drug: Amoxicillin — Group A,Group B,Control group: Amoxicillin capsules 1g, BID, 14days Group D : Amoxicillin capsules 1g, TID, 7 days
  Arms: Control group; Group A; Group B; Group D

SUMMARY:
This is a single-center, randomized, open-label phase Ic/IIb clinical study to evaluate the efficacy and safety of TNP-2198 capsules, rabeprazole sodium enteric-coated tablets and amoxicillin capsules combined with multiple doses of rabeprazole sodium enteric-coated tablets and amoxicillin capsules compared with multiple doses of rabeprazole sodium enteric-coated tablets and amoxicillin capsules combined with multiple doses in Helicobacter pylori infection-positive population.

ELIGIBILITY:
Inclusion Criteria:

* Signing the informed consent form (ICF);
* Male and female subjects aged 18 to 65 years (inclusive);
* Health condition: no clinically significant history of heart, liver, kidney, digestive tract, nervous system, respiratory system diseases, mental disorders or metabolic abnormalities;
* Normal results or clinically insignificant abnormal results in physical examinations and vital signs;
* Positive result of 14C urea breath test (UBT);
* The subject (including the partner) is willing to take effective contraceptive measures voluntarily without pregnancy plan in the next 6 months;
* Willing to follow and able to complete all trial procedures.

Exclusion Criteria:

* History of Helicobacter Pylori eradication therapy (including participation in other clinical studies of Helicobacter Pylori eradication);
* Average daily consumption of more than 5 cigarettes within 3 months prior to the start of the study;
* History of hypersensitivity to study drug or its excipients, or allergic constitution (allergy to multiple drugs and food);
* History of drug and/or alcohol abuse (mean consumption of ≥ 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of liquor, or 100 mL of wine);
* Blood donation or massive blood loss (> 450 mL) within 3 months prior to screening;
* Using any drug that changes liver enzyme activity within 28 days prior to screening;
* Taking orally any prescription drug, over-the-counter drug, any vitamin product, or herbal medicine within 14 days prior to screening;
* Taking special diet (including dragon fruit, mango, grapefruit, etc.) or strenuous exercise, or having other factors that affect drug absorption, distribution, metabolism, excretion, etc., within 2 weeks prior to screening;
* Significant changes in diet or exercise habits recently;
* Those who have participated in, or are still participating in clinical studies within 1 months before taking the study drug;
* With difficulty in swallowing or history of any gastrointestinal diseases that affect drug absorption;
* With any disease that increases the risk of bleeding, such as hemorrhoids, acute gastritis or gastric and duodenal ulcers;
* With clinically significant ECG abnormalities;
* Female subjects who are lactating during the screening period or during the study, or have positive serum pregnancy test results;
* With symptoms or previous history of cardiovascular, digestive, respiratory, urinary, neurological, hematologic, immunological, endocrine system diseases or tumor, or psychiatric diseases;
* Clinically significant abnormalities in clinical laboratory tests, or other clinically significant findings (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, neoplastic, pulmonary, immunological, psychiatric, or cardiovascular disease);
* Those who have positive tests results of viral hepatitis (including hepatitis B and C), HIV antibody, treponema pallidum antibody (additional Rapid Plasma Reagin（RPR）test is required for those with positive treponema pallidum antibody);
* Acute illness occurs or concomitant medication is used from the date of signing the informed consent to the date prior to study medication;
* Consumption of chocolate, any caffeine- or xanthine-containing food or drink within 48 hours prior to taking the study drug;
* Consumption of any alcoholic product within 48 hours prior to taking the study drug;
* Those who have positive test result of urine drug screening or history of drug abuse or drug addiction within the past 5 years;
* Those who have other conditions that, in the opinion of the investigator, make participation in this study inappropriate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-06-26 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: TenNor Clinical Trials, Study Director — TenNor
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Liu Y, Wang M, Gao L, Liu J, Zhang H, Wu M, Chen H, Lou J, Wang J, Chen J, Geng G, Ma Z, Ding Y. Safety, pharmacokinetics, and efficacy of rifasutenizol, a novel dual-targeted antibacterial agent in healthy participants and patients in China with Helicobacter pylori infection: four randomised clinical trials. Lancet Infect Dis. 2024 Jun;24(6):650-664. doi: 10.1016/S1473-3099(24)00003-3. Epub 2024 Feb 12. PMID 38359854

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Rabeprazole sodium enteric-coated tablets 20 mg + amoxicillin capsules 1 g; BID for 14 days
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D | Control Group
Started | 20 | 20 | 10 | 10 | 20
Completed | 19 | 18 | 10 | 10 | 20
Not Completed | 1 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Control Group | Total
Number analyzed (Participants) | 20 | 20 | 10 | 10 | 20 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 10 | 10 | 20 | 80
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (9.84) | 38.1 (8.65) | 35.8 (9.08) | 40.6 (7.03) | 37.6 (10.62) | 38.5 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 6 | 7 | 7 | 40
  Male | 8 | 12 | 4 | 3 | 13 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 20 | 20 | 10 | 10 | 20 | 80
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Eradication Rate of Helicobacter Pylori Infection
Description: Eradication rate of H. pylori is defined as negative urea breath test result.
Time Frame: Group A, B,C,control group: Urea breath test is assessed Day 44~Day 50 after the first dose; Group D: Urea breath test is assessed Day 37~ Day 43 after the first dose
Population: Modified Intent-to-Treat Analysis Set (mITT): Refers to all randomized participants who have 14C UBT performed on Day 28 to 34 after the last dose of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C | Group D | Control Group
Number analyzed (Participants) | 19 | 19 | 10 | 10 | 20
Participants | 18 | 17 | 5 | 10 | 16

ADVERSE EVENTS:
Time Frame: From Day 1 to Day 44 ~ Day 50 after the first dose
Arm/Group | Group A | Group B | Group C | Group D | Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/10 | 0/10 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/10 | 0/10 | 0/20
Other Adverse Events (participants affected / at risk) | 16/20 | 20/20 | 7/10 | 8/10 | 14/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=20) | Group B (N=20) | Group C (N=10) | Group D (N=10) | Control Group (N=20)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5 | 12 | 2 | 3 | 2
Blood albumin decreased (Investigations) | 5 | 5 | 2 | 2 | 2
Neutrophil count decreased (Investigations) | 3 | 3 | 1 | 1 | 2
Blood bilirubin increased (Investigations) | 1 | 3 | 1 | 1 | 3
Aspartate Aminotransferase increased (Investigations) | 1 | 1 | 1 | 1 | 2
Creatinine renal clearance decreased (Investigations) | 2 | 2 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT06076694/Prot_SAP_000.pdf